CLINICAL TRIAL: NCT05038670
Title: Comparison of Patients-reported Outcome After Total Knee Arthroplasty With Use of Bi-cruciate Stabilized and Personalized Implant Design - Randomized Controlled Trial
Brief Title: Journey II vs Persona Knee Systems - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopedics and Rehabilitation, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WarsawMU/persona
Record Dates: First submitted 2021-08-25; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will not be informed which type of prosthesis was used in their particular case.
  Outcomes Assessor, who will be not present during surgery, will not be informed which type of prosthesis was used in particular patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERSONA (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Zimmer Biomet PERSONA system
  Interventions: Device: Total Knee Replacement
- Journey II (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Smith&Nephew Journey II system
  Interventions: Device: Total Knee Replacement

INTERVENTIONS:
Device: Total Knee Replacement — Participant will undergo total knee replacement performed via anterior parapatellar approach with either PERSONA PS or JOURNEY II BCS

SUMMARY:
This study compares and evaluates differences in patient-reported outcome, survivorship and radiological analysis between patients undergoing total knee arthroplasty with use of either Zimmer Biomet PERSONA Posterior Stabilized (PS) system and Smith&Nephew Journey II Bi-Cruciate Stabilized (BCS) system

DETAILED DESCRIPTION:
The aim of this study is to assess patient-reported outcome, survivorship and radiological analysis in patients after total knee arthroplasty, who will undergo the surgery with the use of either Zimmer Biomet PERSONA Posterior Stabilized (PS) system and Smith&Nephew Journey II Bi-Cruciate Stabilized (BCS) system.

To this study 45 consecutive patients undergoing total knee arthroplasty will be recruited to each group. Study protocol is designed as a prospective, blinded, parallel-group, superiority trial, with balanced randomization [1:1]. All participants will be operated in single clinical orthopedic department, by single high-volume surgeon, who performed more than 3000 total knee arthroplasties in his professional career.

Before the surgery patients will fulfill the author's questionnaire concerning their age, height and body mass, level of activity, WOMAC and KOOS scales.

1-day posteoperatively patients will undergo standard computed tomography examination to assess components placement

ELIGIBILITY:
Inclusion Criteria:

* Listed for a primary total knee replacement (TKR) at the Orthopaedic and Rehabilitation Department Medical University of Warsaw
* Indication for the TKR is primary osteoarthritis of the knee joint involving one or more compartments
* Aged 18 or over
* Patient willing to provide full informed consent to the trial

Exclusion Criteria:

* Listed for a single-stage bilateral TKR procedure
* Severe symptoms in the contralateral knee so as to require staged bilateral knee replacements within 6 months of the primary procedure
* Fixed flexion deformity of 15 degrees or greater who will require excessive resection of the distal femur
* Clinically assessed uncorrectable varus/valgus deformity of 15 degrees or greater
* Any co-morbidity which, in the opinion of the investigator, is severe enough to present an unacceptable risk to the patient's safety
* Inflammatory arthritis
* Previous septic arthritis in the affected knee joint
* Previous surgery to the collateral ligaments of the affected knee
* Patients on warfarin or novel oral anticoagulants (NOACs)
* Will not be resident in the catchment area for at least 6 months post-surgery
* Undertaking the surgery as a private patient
* Patients who, in the opinion of the clinical staff, do not have capacity to consent
* Patients who are pregnant
* Unable to understand written and spoken Polish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Changes in patients reported outcome measures - KOOS Score (Knee injury and Osteoarthritis Outcome Score) | baseline (preoperatively) and 1 year postoperatively
  To explore differences between outcome in patients treated with use of with Journey II and Persona prosthesis. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcome measures - WOMAC Score (Knee injury and Osteoarthritis Outcome Score) | baseline (preoperatively) and 1 year postoperatively
  To explore differences between outcome in patients treated with use of with Journey II and Persona prosthesis. Results range from 0 to 96, with higher scores corresponding to worse outcomes.
Values of components rotation | 1-day postoperatively
  Values of external or internal rotation of components measured in computed tomography postoperatively. Values in degrees in regards to anatomic bone landmarks

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolaerczyk, MD, PhD, Principal Investigator — Department of Orthopedics and Rehabilitation, Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes